CLINICAL TRIAL: NCT05093751
Title: Automated Meningioma Segmentation and Volumetry Using a nnU-Net Based Architecture on Contrast-enhanced MRI
Brief Title: Automated Segmentation and Volumetry for Meningioma Using Deep Learning
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chul-Kee Park, Professor, Seoul National University Hospital
Other Study IDs: SNUH-MNG-AI001
Record Dates: First submitted 2021-10-01; First posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Meningioma; Artificial Intelligence
Keywords: Meningioma; Artificial intelligence; autosegmentation; volumetry
MeSH Terms: conditions — Meningioma | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Meningioma patients
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — This study does not involve any intervention to subjects.

SUMMARY:
U-Net-based architectures will be applied to 500 contrast-enhanced axial MR images of different patients from a single institution after manual segmentation of meningioma, of which 50 were used for testing. Tumor volumetry after autosegmentation by trained U-Net-based architecture is final goal.

DETAILED DESCRIPTION:
U-Net-based architectures will be applied to 500 contrast-enhanced axial MR images of different patients from a single institution after manual segmentation of meningioma, of which 50 were used for testing. After preprocessing with Z-isotropification and intensity normalization of images, 3 U-Net-based networks (2D U-Net, Attention U-Net, 3D U-Net) and 3 nnU-Net-based networks (2D nnU-Net, Attention nnU-Net, 3D nnU-Net) will be trained with meningioma-segmented images. For applying to 3D networks, sagittal and coronal images will be reconstructed using axial images. After prediction, the cut-off of the probability function, which is a trade-off, will be obtained with the Gaussian Mixture Modeling algorithm using the probability density function. The voxels having a probability function higher than that will be finally predicted as meningioma. Tumor volume is calculated as the sum of the product of segmented area and thickness of axial images. For performance evaluation, dice similarity coefficient (DSC), precision, and recall will be evaluated compared with manually segmented voxels for validation datasets. The results of volumetry of each model will be compared with manual segmentation-based volume through Pearson's correlation analysis.

ELIGIBILITY:
Inclusion Criteria:

* Radiologically diagnosed meningioma by MRI

Exclusion Criteria:

* under 18 years old
* Multiple meningiomas
* Orbital meningioma
* Any prior treatment for intracranial meningioma before registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intracranial meningioma patients who were diagnosed by MRI are study population of this study. Inclusion in this study have not been decided according to whether or not surgery for tumor resection was performed or MRI thickness and magnetic power.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2013-03-23 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Accuracy compared with ground truth | 10-01-2020 until 09-30-2021
  As a primary endpoint, we will examine the ability of U-Net and nnU-Net to segment meningioma in brain MR compared with ground truth. Ground truth is defined as area on MR drawn by two neurosurgeons. Accuracy of autosegmentation of meningioma will be assessed in dice similarity coefficient, recall, and precision.

IPD SHARING:
Plan to Share IPD: No
We have no plan to share IPD